CLINICAL TRIAL: NCT06377150
Title: ABCA4-associated Disease in Childhood and Adolescence - a Phenotype Study
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: ABCA4-1382022BO2
Record Dates: First submitted 2024-04-12; First posted 2024-04-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-04

CONDITIONS: Stargardt Disease
Keywords: Stargardt Disease; ABCA4; inherited retinal dystrophy
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Retrospective chart review study to elucidate the phenotype and genotype of children with ABCA4-associated Stargardt disease.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed ABCA4-associated inherited retinal dystrophy

Exclusion Criteria:

* 18 years old and older

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with genetically confirmed ABCA4-associated inherited retinal dystrophy.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | January 2014 - May 2021
  best corrected visual acuity
Visual Field (VF) | January 2014 - May 2021
  visual field as measured by semi-automated 90° kinetic visual field exam using target III4e
Fundus Photography (FP) | January 2014 - May 2021
  characterization of the retina with fundus photography
Fundus Autofluorescence (AF) | January 2014 - May 2021
  characterization of the retina with fundus autofluorescence
Optical Coherence Tomography (OCT) | January 2014 - May 2021
  characterization of the retina with optical coherence tomography, e.g. foveal ellipsoid zone loss
Full-Field Electroretinography (ff-ERG) | January 2014 - May 2021
  characterization of retinal function with full-field electroretinogram

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kuehlewein, MD, Principal Investigator — Centre for Ophthalmology, University of Tuebingen; Susanne Kohl, PhD, Principal Investigator — Molecular Genetics Laboratory, Centre for Ophthalmology, University of Tuebingen; Jan-Philipp Bodenbender, MD, Principal Investigator — Centre for Ophthalmology, University of Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wuerttemberg, Germany, Germany

IPD SHARING:
Plan to Share IPD: No